CLINICAL TRIAL: NCT01654406
Title: Fractional CO2 Laser in the Treatment for Cesarian Scar
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: because 1 patient's scar becomes more severe than before, and most patient have satificated outcome
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-JIRB 201203007
Record Dates: First submitted 2012-07-24; First posted 2012-07-31 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Cesarian Scar
Keywords: Cesarian scar; Fractional CO2 laser
MeSH Terms: interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Control (Active Comparator): Pulsed dye laser (V-beam)
  Interventions: Device: Pulsed dye laser
- Experimental group (Experimental): Fractional CO2 laser(eCO2)and pulsed dye laser (V-beam)
  Interventions: Device: Fractional CO2 laser and pulsed dye laser

INTERVENTIONS:
Device: Fractional CO2 laser and pulsed dye laser — Fractional CO2 laser: 50 mJ, 100 spots/cm2, a scan area of 4_4mm, static mode, and two passes Pulsed dye laser: 5mm,1.5ms,8J,delay cooling device 30/30,one pass
  Arms: Experimental group
Device: Pulsed dye laser — Pulsed dye laser: 5mm,1.5ms,8J,delay cooling device 30/30,one pass
  Arms: Control

SUMMARY:
Fractional CO2 laser can improve the Cesarian scar

ELIGIBILITY:
Inclusion Criteria:

* Female receiving Cesarean surgery for more than 1 month

Exclusion Criteria:

* Pregnancy
* Keloid
* Photosensitivity
* Wound
* Pacemaker
* Recent retinoid intake

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
change of Vancouver Scar Scale (VSS) | 1st, 5th, 7th month
  We measured quartile grading scale at 1st, 5th and 7th months of study and evaluated the change of the scale

SECONDARY OUTCOMES:
Quartile grading scale | 5th, 7th month
  We measured quartile grading scale at 5th and 7th months of study.

CONTACTS AND LOCATIONS:
Locations (1):
- Wan Fang Hospital, Taipei, Taiwan, Taiwan